CLINICAL TRIAL: NCT05151991
Title: A 12-months Evaluation of the Failure Rates of Stainless Steel and Ceramic Brackets in Orthodontic Fixed Therapy: a Clinical Trial.
Brief Title: A Clinical Trial on the Failure Rates of Metallic and Ceramic Orthodontic Brackets
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pavia (Other)
Responsible Party: Principal Investigator, Andrea Scribante, Research Resident, Principal Investigator, University of Pavia
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2021-METCERORTO
Record Dates: First submitted 2021-11-10; First posted 2021-12-09 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Dental Malocclusion
Keywords: metallic brackets; ceramic brackets; bond failures; multibrackets therapy; orthodontic treatment; bonding
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Groups MET (Active Comparator): Patients from this group will undergo orthodontic fixed treatment with stainless steel brackets.
  Interventions: Other: Fixed orthodontic treatment with stainless steel brackets
- Group CER (Active Comparator): Patients from this group will undergo orthodontic fixed treatment with ceramic brackets.
  Interventions: Other: Fixed orthodontic treatment with ceramic brackets

INTERVENTIONS:
Other: Fixed orthodontic treatment with stainless steel brackets — Orthophosphoric acid 37% acid (Gerhò Etchant gel 37%, Gerhò spa, Terlano, Italy) will be applied for 30 s for the etching of the vestibular surfaces of teeth. The, after rinsing and drying, a thin layer of Transbond XT Light Cure Adhesive Primer (3M Unitek, Monrovia, CA, USA) will be applied and then cured for 10 s with a LED unit. At last, Transbond XT Light Cure Adhesive Paste (3M Unitek) will be applied on the base of stainless steel brackets (Queen Series Low Profile Brackets MBT 0.022", Aestetika, Terni, TR, Italy); brackets will be applied on the vestibular surfaces of teeth with a light pressure and the extra paste will be removed. Curing will be performed with the LED unit at 2 mm distant from the enamel-bracket interface for 40 s, 10 s per each surface (mesial, distal, gingival and occlusal). The following sequence of archwires will be adopted for the first six months: 0.012-in Niti, 0.014-in Niti, 0.016-in NiTi, 0.018 SS, 0.020 SS, 0.017X0.025-in NiTi, 0.019X0.025-in SS.
  Arms: Groups MET
Other: Fixed orthodontic treatment with ceramic brackets — Orthophosphoric acid 37% acid (Gerhò Etchant gel 37%, Gerhò spa, Terlano, Italy) will be applied for 30 s for the etching of the vestibular surfaces of teeth. The, after rinsing and drying, a thin layer of Transbond XT Light Cure Adhesive Primer (3M Unitek, Monrovia, CA, USA) will be applied and then cured for 10 s with a LED unit. At last, Transbond XT Light Cure Adhesive Paste (3M Unitek) will be applied on the base of ceramic brackets; brackets (Super Clear Series Brackets MBT 0.022", Aestetika, Terni, TR, Italy) will be applied on the vestibular surfaces of teeth with a light pressure and the extra paste is removed. Curing will be performed with the LED unit at 2 mm distant from the enamel-bracket interface for 40 s, 10 s per each surface (mesial, distal, gingival and occlusal). Then, the following sequence of archwires will be adopted for the first six months: 0.012-in Niti, 0.014-in Niti, 0.016-in NiTi, 0.018 SS, 0.020 SS, 0.017X0.025-in NiTi, 0.019X0.025-in SS
  Arms: Group CER

SUMMARY:
The aim of this study is to assess if there are significant differences in the failure rate of stainless steel and ceramic brackets. For this study, patients will be enrolled and divided into two groups, according to the type of brackets (stainless steel or ceramic) used for orthodontic treatment. Failure rates will be recorded every month for 12 months and survival analysis will be performed, together with skeletal and space analysis.

DETAILED DESCRIPTION:
This clinical trial aims to investigate if there are differences in the failure rates of stainless steel and ceramic orthodontic brackets. Patients willing to start orthodontic fixed therapy and recruited for the study will be asked to sign the informed consent. Parents will sign the consent for underage patients. After that, patients will be divided into two groups:

* Group MET: stainless steel brackets will be bonded on the vestibular surfaces of teeth.
* Group CER: ceramic brackets will be bonded on the vestibular surfaces of teeth. The following sequence of archwires will be adopted for the first six months: 0.012-in Niti, 0.014-in Niti, 0.016-in NiTi, 0.018 SS Australian, 0.020 SS Australian, 0.017X0.025-in NiTi, 0.019X0.025-in SS. The failure rates of the brackets will be recorded each month for 12 months. Each failed bracket will be recorded once. For each patient, pre-treatment lateral cephalometric radiograph and study models will be used to measure ANB angle, Wits, Skeletal Class, dento-alveolar discrepancy and Little Index at the beginning of the treatment. Bond failures will be recorded together with the archwire engaged at the moment of the failure.

Sample size Sample size was calculated with the following assumptions: ability to detect a clinically relevant difference of 4.935% in the failure rates (primary outcome) of the two groups with an alfa = 0.05 and power = 80%. The assumptions were based on findings of a previous study with an expected value of 12.08% for the first group at the end of 12 months of therapy. Therefore, 800 brackets (40 patients) per group were required for the study.

Statistical analysis Statistical analysis will be conducted with R software (R version 3.1.3, R Development Core Team, R Foundation for Statistical Computing, Wien, Austria). Fisher exact test will be performed to evaluate the differences between the failure rates of the two groups, between anterior and posterior sites and between upper and lower arches. Kaplan-Meier survival analysis of the bond failures will be performed among the 12 months of the study. Linear regressions will be calculated to assess the effects on bond failure of the skeletal and dental variables collected before the bonding procedure. Significance for all statistical tests will be predetermined at P<0.05.

ELIGIBILITY:
Inclusion Criteria:

* patients willing to begin fixed multibracket therapy with metallic or ceramic brackets;
* full permanent dentition;
* enamel integrity, absence of traumatic or carious lesions, no pretreatment procedure performed with chemical agents;
* no previous orthodontic treatment with fixed vestibular appliances.

Exclusion Criteria:

* patients suffering from systemic diseases;
* patients taking medications that could alter periodontal conditions (NSAIDS, steroids, etc.);
* patients with low compliance;
* patients unable to give informed consent;
* presence of congenital enamel defects;
* extractions for orthodontic reasons;
* oral/orthognathic surgery.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-12-09 (Actual); Primary Completion 2023-05-04 (Actual); Study Completion 2023-05-08 (Actual)

PRIMARY OUTCOMES:
Failure rates of metallic and ceramic brackets. | Among the 12 months of the study.
  Each month, failed brackets will be recorded. Per each tooth, failure will be recorded once.

SECONDARY OUTCOMES:
Failure rates of metallic and ceramic brackets per sites and sides. | Among the 12 months of the study.
  Failures will be divided in "anterior" for brackets failed on incisors and canines, and "posterior" for premolar brackets. Failure will be recorded per dental arch ("upper" and "lower") and per archwire (.014-in NiTi, .016-in NiTi, .017X0.25-in NiTi, .019X.025-in SS). Per each tooth, failure will be recorded once.
ANB angle | Before the beginning of the orthodontic treatment.
  ANB angle will be calculated using the pre-treatment lateral cephalometric radiograph.
Wits Index | Before the beginning of the orthodontic treatment.
  Wits Index will be calculated using the pre-treatment lateral cephalometric radiograph.
Skeletal Class | Before the beginning of the orthodontic treatment.
  Skeletal Class will be assessed using ANB angle and Wits Index will be calculated using the pre-treatment lateral cephalometric radiograph.
Dento-alveolar discrepancy | Before the beginning of the orthodontic treatment.
  Dento-alveolar discrepancy will be calculated using the pre-treatment study models.
Little Index | Before the beginning of the orthodontic treatment.
  Little Index will be calculated using the pre-treatment study models.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Scribante, DDS, PhD, Principal Investigator — University of Pavia
Locations (1):
- Unit of Orthodontics and Pediatric Dentistry - Section of Dentistry - Department of Clinical, Surgical, Diagnostic and Pediatrics - University of Pavia, Pavia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No
Data will be available upon motivated request to Principal Investigator

REFERENCES:
- [Background] Kirschneck C, Rohn C, Proff P, Reicheneder C. Influence of enamel sealing with a light-cured filled sealant before bracket bonding on the bond failure rate during fixed orthodontic therapy. J Orofac Orthop. 2019 May;80(3):136-143. doi: 10.1007/s00056-019-00174-w. Epub 2019 Apr 10. PMID 30972424